CLINICAL TRIAL: NCT02228070
Title: Strabismus Measurements Using Automated 3D Video Oculography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Albert Bruppacher-Stiftung (Unknown); Stiftung OPOS zugunsten von Wahrnehmungsbehinderten (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK-ZH-Nr. 2014-0481
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Strabismus
Keywords: strabismus; oculomotor palsy; abducens palsy; trochlear palsy
MeSH Terms: conditions — Strabismus; Abducens Nerve Diseases

ARMS (1):
- strabismus video goggles (Experimental)
  Interventions: Device: strabismus video goggles

INTERVENTIONS:
Device: strabismus video goggles

SUMMARY:
Measuring ocular motility and alignment is important for diagnosing different causes of strabismus, following patients recovering from cranial nerve palsies, preparing patients for strabismus surgery and follow-up post surgery. The current clinical gold standards for measuring ocular alignment are the Hess screen and the Harms tangent screen. These tests are accurate, but require patient cooperation, and are not objective because the patient has to indicate the position of the light he sees on the screen. Our objective is to develop an accurate and easy to use goggles system to measure ocular alignment and motility using 3D video oculography.

ELIGIBILITY:
Inclusion Criteria:

* Patients 11 years or older
* congenital strabismus
* acquired strabismus
* paretic strabismus (oculomotor, abducens and trochlear nerves)
* before and after strabismus surgery
* normal controls

Exclusion Criteria:

* Patients unable to sign informed consent
* Patients with significantly impaired vision
* Patients unable to cooperate with standard strabismus workup (including Hess and Harms tests)
* For sub-study: intolerance to scleral search coils

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Validation of video goggles against Hess/Harms screen | initial visit
  Measurement of squint angle with 3D video goggles vs. Hess/Harms screen.

SECONDARY OUTCOMES:
Accuracy of video goggles in comparison to scleral search coils | initial visit
  Measurement of squint angle with 3D video goggles vs. scleral search coils.

OTHER OUTCOMES:
Follow-up squint angle measures post-OP and after recovery from cranial nerve palsy with 3D video goggles and Hess/Harms screen | initial visit, 3 months after surgery, recovery from cranial nerve palsy after 3 months
  Change in squint angle with 3D video goggles and Hess/Harms screen.

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology Department, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Weber KP, Rappoport D, Dysli M, Schmuckle Meier T, Marks GB, Bockisch CJ, Landau K, MacDougall HG. Strabismus Measurements with Novel Video Goggles. Ophthalmology. 2017 Dec;124(12):1849-1856. doi: 10.1016/j.ophtha.2017.06.020. Epub 2017 Jul 17. PMID 28728924